CLINICAL TRIAL: NCT06328036
Title: Phase 2 and Biomarker Trial of Anti-TIGIT and Anti-PDL1 in Patients With Recurrent Glioblastoma
Brief Title: Testing the Combination of Anti-cancer Drugs Tiragolumab and Atezolizumab to Improve Outcomes for Patients With Recurrent Glioblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - Protocol moved to Disapproved
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-02185; NCI-2024-02185 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10640 (Other: UPMC Hillman Cancer Center LAO); 10640 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-03-25 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Glioblastoma, IDH-Wildtype
MeSH Terms: conditions — Glioblastoma | interventions — atezolizumab; Specimen Handling; Magnetic Resonance Spectroscopy; Surgical Procedures, Operative; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- GROUP A (neoadjuvant atezolizumab, tiragolumab) (Experimental): Patients receive atezolizumab IV over 60 minutes and tiragolumab IV over 20-75 minutes and 14-19 days later, undergo surgical resection. Following surgery, patients may receive tiragolumab IV and atezolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI at baseline, 24-72 hours after surgery, then every 9 weeks until progression and blood sample collection throughout the study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Procedure: Surgical Procedure; Biological: Tiragolumab
- GROUP B (neoadjuvant tiragolumab) (Experimental): Patients receive tiragolumab IV over 20-75 minutes and 14-19 days later, undergo surgical resection. Following surgery, patients may receive tiragolumab IV and atezolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI at baseline, 24-72 hours after surgery, then every 9 weeks until progression and blood sample collection throughout the study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Procedure: Surgical Procedure; Biological: Tiragolumab
- GROUP C (neoadjuvant atezolizumab) (Experimental): Patients receive atezolizumab IV over 60 minutes and 14-19 days later, undergo surgical resection. Following surgery patients may receive atezolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI at baseline, 24-72 hours after surgery, then every 9 weeks until progression and blood sample collection throughout the study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Procedure: Surgical Procedure
- GROUP D (no neoadjuvant drug) (Active Comparator): Patients undergo surgical resection on study. Following surgery patients may receive atezolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI at baseline, 24-72 hours after surgery, then every 9 weeks until progression and blood sample collection throughout the study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Procedure: Surgical Procedure; Biological: Tiragolumab

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Surgical Procedure — Undergo surgical resection
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
Biological: Tiragolumab — Given IV
  Other Names: MTIG7192A; RG6058
  Arms: GROUP A (neoadjuvant atezolizumab, tiragolumab); GROUP B (neoadjuvant tiragolumab); GROUP D (no neoadjuvant drug)

SUMMARY:
This phase II trial compares the safety, side effects and effectiveness of atezolizumab with tiragolumab to atezolizumab alone in treating patients with glioblastoma that has come back after a period of improvement (recurrent). Glioblastoma is the most common primary brain cancer in adults and despite aggressive treatment, it is nearly always fatal. Currently, there are limited effective treatment options in patients that have recurrence. Immunotherapy has been shown to be effective in other types of cancer and may be an appealing potential treatment option for recurrent glioblastoma. Immunotherapy with monoclonal antibodies, such as atezolizumab and tiragolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Study doctors also want to learn if a tumor infiltrating T lymphocyte (TIL) response is helpful to determine the benefit of the combination of study drugs compared to the usual approach. TILs are a type of immune cell that has moved from the blood into a tumor. TILs can recognize and kill tumor cells. Giving atezolizumab with tiragolumab may be safe, tolerable and/or effective compared to atezolizumab alone in treating patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the impact of combination atezolizumab plus tiragolumab on progression free survival.

SECONDARY OBJECTIVES:

I. To evaluate the impact of atezolizumab, tiragolumab, or their combination on tumor infiltrating T lymphocyte (TIL) density in glioblastoma patients.

II. To evaluate the safety of study drug therapy in patients with glioblastoma in the (neo)adjuvant setting.

III. To estimate therapeutic benefit of atezolizumab and tiragolumab in the recurrent glioblastoma patient population.

IV. To evaluate the impact of baseline tumor mutation burden and expression on response.

EXPLORATORY OBJECTIVES:

I. To evaluate the impact of combination treatment on the tumor immune microenvironment.

II. To evaluate the impact of combination treatment on the peripheral immune microenvironment.

III. To evaluate the peripheral and central pharmacokinetics of tiragolumab and atezolizumab.

OUTLINE: Patients are randomized to 1 of 4 groups.

GROUP A: Patients receive atezolizumab intravenously (IV) over 60 minutes and tiragolumab IV over 20-75 minutes and 14-19 days later, undergo surgical resection. Following surgery, patients may receive tiragolumab IV and atezolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo magnetic resonance imaging (MRI) at baseline, 24-72 hours after surgery, then every 9 weeks until progression and blood sample collection throughout the study.

GROUP B: Patients receive tiragolumab IV over 20-75 minutes and 14-19 days later, undergo surgical resection. Following surgery, patients may receive tiragolumab IV and atezolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI at baseline, 24-72 hours after surgery, then every 9 weeks until progression and blood sample collection throughout the study.

GROUP C: Patients receive atezolizumab IV over 60 minutes and 14-19 days later, undergo surgical resection. Following surgery patients may receive atezolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI at baseline, 24-72 hours after surgery, then every 9 weeks until progression and blood sample collection throughout the study.

GROUP D: Patients undergo surgical resection on study. Following surgery patients may receive atezolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI at baseline, 24-72 hours after surgery, then every 9 weeks until progression and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed IDH wildtype World Health Organization (WHO) grade IV glioblastoma at first or second relapse
* Documented progression of disease as defined by modified Response Assessment in Neuro-Oncology (mRANO) criteria at least 12 weeks after completion of radiotherapy, unless the recurrence is outside the radiation field or has been histologically documented
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of atezolizumab in combination with tiragolumab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky ≥ 60%)
* Leukocytes ≥ 2,000/mcL
* Lymphocyte count ≥ 500/mcL
* Absolute neutrophil count ≥ 1,500/mcL without granulocyte colony-stimulating factor support
* Platelets ≥ 100,000/mcL without transfusion
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x institutional ULN or ≤ 5 x ULN for patients with liver metastases
* Alkaline phosphatase ≤ 2.5 x ULN (≤ 5 x ULN for patients with documented liver or bone metastases)
* Glomerular filtration rate (GFR) ≥ 30 mL/min
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN (This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-weight heparin or warfarin, should be on a stable dose.)
* Serum albumin ≥ 2.5 g/dL
* Negative human immunodeficiency virus (HIV) test at screening with the following exception: individuals with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4+ T cell count ≥ 200/uL, and have an undetectable viral load
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following:

  * Negative total hepatitis B core antibody (HBcAb)
  * Positive total HBcAb test followed by quantitative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) < 500 IU/mL. The HBV DNA test will be performed only for patients who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients must be undergoing surgery that is clinically indicated as determined by their care providers
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with IDH mutations will be excluded from the study
* Patients who have had previous treatment with anti PD1, PDL1, CTLA-4 or other immune checkpoint inhibitors
* Patients who have undergone tumor directed therapy for the most recent disease progression
* Patients who have not recovered to grade 0 or 1 or pre-treatment baseline from clinically significant adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients with a diagnosis of immunodeficiency or who require treatment with high dose systemic corticosteroids defined as dexamethasone > 2 mg/day or bioequivalent for at least 3 consecutive days within 1 week of start of study drug
* Patients with severe, uncontrolled intercurrent illness, comorbidity, or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Patients who are pregnant or breastfeeding or are expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 5 months after the last dose of study treatment. Women of childbearing potential (WOCPB) must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment. A WOCBP who has a positive urine pregnancy test (e.g., within 72 hours) prior to treatment will be excluded from the study. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Per this definition, a woman with a tubal ligation is considered to be of childbearing potential. The definition of childbearing potential may be adapted for alignment with local guidelines or regulations. Pregnant women are excluded from this study because atezolizumab and tiragolumab are monoclonal antibodies with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with atezolizumab and/or tiragolumab, breastfeeding should be discontinued if the mother is treated with atezolizumab and/or tiragolumab. To avoid pregnancy, WOCBPs and men must agree to use adequate contraception (i.e., contraceptive methods with a failure rate of < 1% per year such as bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices) prior to the study, during treatment, and for 5 months after treatment ends. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patients unable to comply with the protocol and/or not willing or who will not be available for follow-up assessments, specifically MRI scans
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the exceptions listed below:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study
  * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-alpha [TNF-alpha] agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
* Patients with presence of extracranial metastatic or leptomeningeal disease
* Patients that have received anti-angiogenic or anti-VEGF targeted agents (e.g., bevacizumab, cediranib, aflibercept, vandetanib, XL-184, sunitinib, etc.)
* Patients with patent active tuberculosis (TB)
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Patients being treated with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 4 weeks prior to cycle 1, day 1. The study principal investigator (PI) must be consulted if a patient was being treated with any antibody within 4 half-lives of said antibody
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis
* Patients treated with therapeutic oral (PO) or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX®) are allowed
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Uncontrolled tumor-related pain:

  * Patients requiring pain medication must be on a stable regimen at study entry
  * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period
  * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural compression) should be considered for loco-regional therapy if appropriate prior to enrollment
* Significant cardiovascular disease (such as New York Heart Association class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrythmia, or unstable angina
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment, within 90 days after the final dose of tiragolumab, or within 5 months after the final dose of atezolizumab
* Positive Epstein-Barr virus (EBV) viral capsid antigen immunoglobulin M (IgM) test at screening. An EBV polymerase chain reaction (PCR) test should be performed as clinically indicated to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or tiragolumab formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 36 months
  Will be assessed and compared between adjuvant arms. PFS will be assessed using Kaplan-Meier method.

SECONDARY OUTCOMES:
Tumor infiltrating T lymphocyte density | Up to 36 months
  Will be assessed and compared between arms. The number of T cells/nucleated cells will be quantified in each sample and the density will be estimated between each treatment group.
Dose limiting toxicity | Up to 30 completion of adjuvant cycle 2
  Will be defined as any grade ≥ 3 non-hematologic toxicity despite best supportive care or grade ≥ 4 hematologic toxicity per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 attributed as possibly, probably, or definitely related to therapy.
Incidence of adverse events | Up to 30 days after last dose of study treatment
  Will be tabulated using CTCAE v 5.0 grading criteria.
Objective response rate (ORR) | Up to 36 months
  Will be assessed based on modified Response Assessment in Neuro-Oncology. ORR will be defined as the summation of complete response and partial response. The probability of ORR will be estimated with exact 95% binomial confidence intervals.
PFS6 | At 6 months
  Will be estimated with exact 95% binomial confidence intervals.
Overall survival | Up to 36 months
  Will be estimated by the Kaplan-Meier method with log rank test, along with 95% confidence regions.
Tumor mutational burden (TMB) | Up to 36 months
  Will be evaluated in each patient and correlation assessment will be performed between T-cell density, gene response set values and other secondary endpoints by Spearman's correlation coefficient.
Expression of immune checkpoint receptors and ligands | Up to 36 months
  Expression of immune checkpoint receptors and ligands will be evaluated. Expression levels will be evaluated in each patient and correlation assessment will be performed between T-cell density, gene response set values and other secondary endpoints by Spearman's correlation coefficient.

OTHER OUTCOMES:
Tumor response signatures including for T-cells, interferon and cell cycle | Up to 36 months
  The statistical differences between groups A, B, C versus (vs) A vs B and C for each gene set will be compared using a non-parametric paired test, at a significance level (alpha) of 0.05 uncorrected for multiple testing.
T cell receptor (TCR) clonality and diversity | Up to 36 months
  The statistical differences between groups A, B, C vs D and A vs B and C fore each gene set will be compared using a non-parametric paired test, at a significance level of 0.05 uncorrected for multiple testing.
Tumor infiltrating T-cell, T-regs, and myeloid cells | Up to 36 months
  Specific immune cell populations and ratios in tumor tissue will be compared between the groups using a non-parametric test, at a significance level of 0.05 uncorrected for multiple testing.
TCR overlap and clonal expression | Up to 36 months
  TCR clones will be evaluated by ImmunoSEQA. Percentage of TCR overlap between tumor tissue and blood at the time of surgery will be calculated for each patient and compared between the groups by non-parametric tests at a significance level of 0.05. Total numbers of clonall expanded T-cells will also be assessed.
Peripheral blood mononuclear cell (PBMC) response signatures including for T-cells, interferon and cell cycle | Up to 36 months
  After correction for batch effect gene set variation analysis scores for each gene set described will be calculated for each patient tumor sample. The statistical difference between groups A, B, C vs D and A vs B and C for each gene set will be compared using a non-parametric paired test, at a significance level (alpha) of 0.05 uncorrected for multiple testing.
TCR clonality by PBMC | Up to 36 months
  Unique T-cell clones, and changes in TCR clone frequencies will be followed through treatment and will be compared between the groups and changes within each patient over time from baseline to each blood draw with a non-parametric tests, (paired within patients; unpaired between groups) at a significance level (alpha) of 0.05.
TCR clonality | Up to 36 months
  A percentage of TCR overlap between tumor tissue and blood at the time of surgery will be calculated for each patient and compared between the groups by non-parametric tests at a significance level of 0.05. Additional assessments will include total numbers of clonally expanded T-cells (> 3 cells sharing a TCR) within a patient.
Trough concentrations in serum and concentrations in cerebrospinal fluid | Up to 36 months
  Pharmacokinetics exposure values will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Mantica, Principal Investigator — University of Pittsburgh Cancer Institute LAO

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm